CLINICAL TRIAL: NCT03694353
Title: An Open-label Extension Study to Evaluate the Safety and Efficacy of Subcutaneous Injections of Pegvaliase (> 40 mg/Day Dose) in Adults With Phenylketonuria
Brief Title: Safety and Efficacy of Self Administered Injections of Pegvaliase (>40mg/Day Dose) in Adults With PKU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 165-304
Record Dates: First submitted 2018-09-04; First posted 2018-10-03 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegvaliase (Experimental): Beginning on Day 1, subjects will receive the same dose and regimen of pegvaliase they were receiving in 165-302 or PAL-003 (pegvaliase dosing should continue without interruption from the previous study). Subsequent revisions to dosing regimens are allowed following consultation with the medical monitor.
  Interventions: Drug: Pegvaliase

INTERVENTIONS:
Drug: Pegvaliase — 40-60mg/day
  Other Names: rAvPAL-PEG

SUMMARY:
This is a Phase 3 open-label extension study enrolling adult patients with PKU who were previously treated with pegvaliase in Studies PAL-003 (NCT00924703) or 165-302 (NCT02468570). The study is designed to evaluate the long-term safety and efficacy of pegvaliase administered at doses > 40 mg/day to 60 mg/day.

DETAILED DESCRIPTION:
Pegvaliase dosing will continue without interruption from Parent Study 165-302 (NCT02468570) or Parent Study PAL-003 (NCT00924703). Beginning on Day 1, subjects will receive the same dose and regimen of pegvaliase they were receiving in either 165-302 or PAL-003. A subject who reduces to a dose of 40 mg/day or lower for 32 consecutive weeks will be discontinued from study drug and withdrawn from the study as they will have the option to transition to commercial drug. Dose reductions may be performed if warranted due to AEs or hypophenylalaninemia. Dose increases to up to 60 mg/day may be performed per investigator discretion in consultation with the sponsor's medical monitor. Dosing will continue for approximately 121 weeks.

ELIGIBILITY:
Inclusion criteria:

* Must be enrolled in PAL-003 or 165-302 Part 4 at the time of screening for 165-304 and most recently receiving pegvaliase at a dose > 40 mg/day.
* Has identified a competent person or persons ≥ 18 years of age who can observe the subject during study drug administration and for a minimum of 1 hour following administration in situations required per protocol.
* For females with childbearing potential, must have negative pregnancy test at screening and be willing to have additional pregnancy tests during the study.
* If sexually active and not planning to become pregnant (self or partner), must be willing to use 2 acceptable methods of contraception while participating in the study and for 4 weeks after the study.
* Is willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures; a legally authorized representative may provide written consent and assent may be requested.
* Is willing and able to comply with all study procedures.
* Is in generally good health, as evidenced by physical examination and/or clinical laboratory evaluations (hematology, chemistry, and urinalysis).

Exclusion criteria:

* Use of any investigational product (except pegvaliase) or investigational medical device within 30 days prior to screening or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Use of any medication (except pegvaliase) intended to treat PKU, including the use of large neutral amino acids, within 2 days prior to the administration of pegvaliase (Day 1).
* Use or planned use of any injectable drugs containing PEG (other than pegvaliase), including medroxyprogesterone injection, within 3 months prior to screening and during study participation.
* A history of organ transplantation or on chronic immunosuppressive therapy
* A history of substance abuse (as defined by the American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders [DSM]) in the past 12 months or current alcohol or drug abuse
* Current participation in the Kuvan® registry study (PKU Demographics, Outcomes and Safety [PKUDOS])
* Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease)
* Any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or terminating early from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (17):
- United States (17):
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Wayne State University, Center for Molecular Medicine and Genetics, Pediatrics and Pathology, Detroit, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Medical College of Milwaukee, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study, conducted in 17 study centers in the United States involving subjects from either Parent Study 165-302 (NCT02468570) or Parent Study PAL-003 (NCT00924703).
Groups:
- All Subjects: Self administered subcutaneous pegvaliase injection using a prefilled syringe.
Period: Overall Study
Arm/Group | All Subjects
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Subject received <= 40 mg/day for > 32 weeks | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  years | 28.84 (9.02)
Age, Customized [Count of Participants; unit: Participants] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  Participants
    16 to < 18 years | 2
    Between 18 and < 66 years | 35
    >/= 66 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  Participants
    Female | 15
    Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 36
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 36
    More than one race | 1
    Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  kg | 94.9 (29.75)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  kg/m^2 | 32 (8.41)
Baseline Blood Phe [Mean (Standard Deviation); unit: umol/L] — Parent Study Baseline (i.e., naïve/pretreatment baseline).
  umol/L | 1376.9 (289.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0
Description: A treatment-emergent AE was defined as any adverse event (AE) newly appearing or worsened in severity following initiation of study drug until 4 weeks after last dose of pegvaliase
Time Frame: Up to Day 741 (approximately Week 106)
Population: Population consisted of all subjects receiving at least one dose of pegvaliase during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 37
Participants
  TEAE | 36
  Related TEAE | 17
  Serious TEAE | 7
  Related Serious TEAE | 1

2. Primary Outcome: Change in Blood Phe Concentration
Description: Change in blood phenylalanine (Phe) concentration from Parent Study baseline (naïve/pretreatment).
Time Frame: The Outcome Measure Data Table below uses the 'analysis visit' as defined by the mapping rule in the SAP. The last Phe measurement was mapped to 'analysis visit' week 121. The actual date of the last Phe measurement was day 836 (approximately Week 119).
Population: Efficacy population consisted of all subjects receiving at least one dose of pegvaliase during the study and having a post-treatment blood Phe concentration measurement.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | All Subjects
Number analyzed (Participants) | 37
µmol/L
  Parent Study Baseline (naïve/pretreatment) | 1376.9 (289.77)
  Change from Baseline to Screening/Day 1: number analyzed (Participants) | 30
  Change from Baseline to Screening/Day 1 | -761 (506.7)
  Change from Baseline at week 9 | -970.6 (513.6)
  Change from Baseline at Week 17 | -963.4 (454)
  Change from Baseline at Week 25: number analyzed (Participants) | 33
  Change from Baseline at Week 25 | -830.6 (599.8)
  Change from Baseline at Week 33: number analyzed (Participants) | 35
  Change from Baseline at Week 33 | -999.8 (528)
  Change from Baseline at Week 41: number analyzed (Participants) | 36
  Change from Baseline at Week 41 | -984.1 (545.6)
  Change from Baseline at Week 49: number analyzed (Participants) | 33
  Change from Baseline at Week 49 | -1001.7 (518.3)
  Change from Baseline at Week 57: number analyzed (Participants) | 33
  Change from Baseline at Week 57 | -867 (569.2)
  Change from Baseline at Week 65: number analyzed (Participants) | 25
  Change from Baseline at Week 65 | -913.2 (445)
  Change from Baseline at Week 73: number analyzed (Participants) | 13
  Change from Baseline at Week 73 | -896 (582.8)
  Change from Baseline at Week 81: number analyzed (Participants) | 26
  Change from Baseline at Week 81 | -847.8 (504)
  Change from Baseline at Week 89: number analyzed (Participants) | 26
  Change from Baseline at Week 89 | -962.3 (482.6)
  Change from Baseline at Week 97: number analyzed (Participants) | 27
  Change from Baseline at Week 97 | -865.6 (567.4)
  Change from Baseline at Week 105: number analyzed (Participants) | 18
  Change from Baseline at Week 105 | -817.4 (584.9)
  Change from Baseline at Week 113: number analyzed (Participants) | 2
  Change from Baseline at Week 113 | -1319 (123)
  Change from Baseline at Week 121: number analyzed (Participants) | 1
  Change from Baseline at Week 121 | -1123 (NA) — Only one subject at Week 121 therefore standard deviation is not applicable.

ADVERSE EVENTS:
Time Frame: Up to Day 741 (approximately Week 106)
Description: Only treatment-emergent AEs that occurred and were reported during the study period were included in AE summaries. The incidence, exposure-adjusted event rate, severity grade (assessed per CTCAE version 5.0), and relationship to study drug (per Investigator) for all treatment-emergent AEs were summarized. For AEs occurring more than once during the study, maximum severity was used to summarize AEs by severity.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 7/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=37)
COVID-19 (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=37)
Nasopharyngitis (Infections and infestations) | 13
Influenza (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Helicobacter infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Injection site bruising (General disorders) | 6
Fatigue (General disorders) | 5
Injection site induration (General disorders) | 5
Injection site reaction (General disorders) | 4
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Induration (General disorders) | 2
Injection site erythema (General disorders) | 2
Injection site pain (General disorders) | 2
Injection site pruritus (General disorders) | 2
Pain (General disorders) | 2
Headache (Nervous system disorders) | 12
Migraine (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Sinus headache (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Limb injury (Injury, poisoning and procedural complications) | 5
Contusion (Injury, poisoning and procedural complications) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Amino acid level decreased (Investigations) | 7
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Seasonal allergy (Immune system disorders) | 5
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03694353/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03694353/SAP_001.pdf